CLINICAL TRIAL: NCT01592552
Title: A Multi-Center Longitudinal Biorepository Study to Provide Biospecimens & Clinical Data From Neurological Disease Patients To Approved Pre-Clinical And Clinical Investigators for Drug & Biomarker Studies
Brief Title: A Biospecimen and Clinical Data Study on Patients for Drug & Biomarker Discovery
Status: Completed | Type: Observational
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-ND-01
Record Dates: First submitted 2011-11-16; First posted 2012-05-07 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease; Multiple Sclerosis; Parkinson's Disease; Huntington's Disease; Amyotrophic Lateral Sclerosis (ALS)
Keywords: Alzheimer's Disease; Multiple Sclerosis; Parkinson's Disease; Huntington's Disease; Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Alzheimer Disease; Multiple Sclerosis; Parkinson Disease; Huntington Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Neurological Condition: Collect blood and other biospecimens like saliva, urine and CSF for research purposes.
- Control: Collect blood and other biospecimens like saliva, urine and CSF for research purposes.

SUMMARY:
The purpose of this research project is to collect and store blood samples and clinical data. Researchers can then use the stored samples in future studies. Through such studies, they hope to find new ways to detect, treat, and maybe even prevent or cure health problems.

DETAILED DESCRIPTION:
Blood samples are collected in the comfort and safety of your home by a certified medical professional. We have mobile phlebotomists located in major metropolitan areas around the nation for your convenience.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 to 100 years old
* A diagnosis of neurological condition
* Proof of diagnosis can be provided

Control group: Healthy donors, males and females, 18 to 100 years of age

Exclusion Criteria

* Receipt of blood products within 30 days of study enrollment
* Receipt of an investigational (unapproved) drug within 30 days of study enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A diagnosis of Multiple Sclerosis, Alzheimer's, Huntington's, or Parkinson's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Biospecimens & Clinical Data collection from patients with neurological diseases. | 2 years
  The purpose of this research project is to collect and store blood samples and clinical data. Researchers can then use the stored samples in future studies. Through such studies, they hope to find new ways to detect, treat, and maybe even prevent or cure health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Phil Silkoff, MD, Principal Investigator — Sanguine Biosciences
Locations (1):
- Sanguine Biosciences, Sherman Oaks, California, United States